CLINICAL TRIAL: NCT07085689
Title: Evaluation of the Effectiveness of Various Desensitizing Treatment Protocols in Permanent Teeth Affected by Molar Incisor Hypomineralization
Brief Title: Evaluation of the Effectiveness of Various Desensitizing Treatment Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Beste Ozgur, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUDHF-MIH-desensitization
Record Dates: First submitted 2025-06-23; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-06

CONDITIONS: Molar Incisor Hypomineralization
Keywords: molar incisor hypomineralization; hypersensitivity; desensitization
MeSH Terms: conditions — Molar Hypomineralization; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: four intervention groups, randomized, single-blind clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: All sensitivity assessments were performed blindly by a researcher who did not know the baseline scores or the treatment administered.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 5% Sodium Fluoride Varnish (Active Comparator): After isolating and drying the teeth to be treated using cotton rolls, 5% sodium fluoride (NaF) varnish (Proshield Varnish, President Dental, Munich, Germany) was applied to the tooth surfaces in two thin layers with the help of a disposable microbrush. The cotton rolls were then removed to allow the varnish to come into contact with saliva and harden. After the procedure, participants were advised to avoid consuming hard foods and brushing their teeth for 4 to 6 hours.
  Interventions: Device: Sodium Fluoride Varnish (5%)
- Silver Diamine Fluoride (Active Comparator): After isolating and drying the teeth to be treated using cotton rolls, a gingival barrier (Top Dam, FGM Dental Group, Brazil) was applied around the cervical area of the crown to cover the surrounding gingiva and was light-cured. After applying petroleum jelly to the lips for isolation, the first step, 38% silver diamine fluoride (Riva Star, SDI, Bayswater, Australia), was applied to the entire tooth surface using a disposable microbrush. Immediately afterward, the second step, potassium iodide, was applied generously to the entire tooth surface using another disposable microbrush. The agent was applied until the creamy white appearance on the tooth disappeared. Excess material on the tooth surface was gently dabbed dry with a cotton pellet.
  Interventions: Device: Silver diamine fluoride- potassium iodide
- Aqueous Silver Fluoride (Active Comparator): After isolating and drying the teeth to be treated using cotton rolls, a gingival barrier (Top Dam, FGM Dental Group, Brazil) was applied around the cervical area of the crown to cover the surrounding gingiva and was light-cured. After applying petroleum jelly to the lips for isolation, the first step, 38% aqueous silver fluoride (Riva Star Aqua, SDI, Bayswater, Australia), was applied to the entire tooth surface using a disposable microbrush. Immediately afterward, the second step, potassium iodide, was applied generously to the entire tooth surface using another disposable microbrush. The agent was applied until the creamy white appearance on the tooth disappeared. Excess material on the tooth surface was gently dabbed dry with a cotton pellet.
  Interventions: Device: Aqueous Silver Fluoride
- Hydroxyethyl Methacrylate and Glutaraldehyde (Gluma) (Active Comparator): After isolating and drying the teeth to be treated using cotton rolls, a gingival barrier (Top Dam, FGM Dental Group, Brazil) was applied around the cervical area of the crown to cover the surrounding gingiva and was light-cured. One to two drops of a desensitizing agent containing hydroxyethyl methacrylate and glutaraldehyde (Gluma, Heraeus Kulzer GmbH, Hanau, Germany) were applied to the tooth surface using a disposable microbrush in a rubbing motion. After waiting for 30-60 seconds, the tooth surface was completely dried until the liquid disappeared and the surface lost its shine, and then rinsed with water.
  Interventions: Device: Hydroxyethyl Methacrylate and Glutaraldehyde

INTERVENTIONS:
Device: Sodium Fluoride Varnish (5%) — After isolating and drying the teeth to be treated using cotton rolls, 5% sodium fluoride (NaF) varnish (Proshield Varnish, President Dental, Munich, Germany) was applied to the tooth surfaces in two thin layers with the help of a disposable microbrush. The cotton rolls were then removed to allow the varnish to come into contact with saliva and harden. After the procedure, participants were advised to avoid consuming hard foods and brushing their teeth for 4 to 6 hours.
  Other Names: Proshield Varnish
  Arms: 5% Sodium Fluoride Varnish
Device: Silver diamine fluoride- potassium iodide — After isolating and drying the teeth to be treated using cotton rolls, a gingival barrier (Top Dam, FGM Dental Group, Brazil) was applied around the cervical area of the crown to cover the surrounding gingiva and was light-cured. After applying petroleum jelly to the lips for isolation, the first step, 38% silver diamine fluoride (Riva Star, SDI, Bayswater, Australia), was applied to the entire tooth surface using a disposable microbrush. Immediately afterward, the second step, potassium iodide, was applied generously to the entire tooth surface using another disposable microbrush. The agent was applied until the creamy white appearance on the tooth disappeared. Excess material on the tooth surface was gently dabbed dry with a cotton pellet.
  Other Names: Riva Star
  Arms: Silver Diamine Fluoride
Device: Aqueous Silver Fluoride — After isolating and drying the teeth to be treated using cotton rolls, a gingival barrier (Top Dam, FGM Dental Group, Brazil) was applied around the cervical area of the crown to cover the surrounding gingiva and was light-cured. After applying petroleum jelly to the lips for isolation, the first step, 38% aqueous silver fluoride (Riva Star Aqua, SDI, Bayswater, Australia), was applied to the entire tooth surface using a disposable microbrush. Immediately afterward, the second step, potassium iodide, was applied generously to the entire tooth surface using another disposable microbrush. The agent was applied until the creamy white appearance on the tooth disappeared. Excess material on the tooth surface was gently dabbed dry with a cotton pellet.
  Other Names: Riva Star Aqua
  Arms: Aqueous Silver Fluoride
Device: Hydroxyethyl Methacrylate and Glutaraldehyde — After isolating and drying the teeth to be treated using cotton rolls, a gingival barrier (Top Dam, FGM Dental Group, Brazil) was applied around the cervical area of the crown to cover the surrounding gingiva and was light-cured. One to two drops of a desensitizing agent containing hydroxyethyl methacrylate and glutaraldehyde (Gluma, Heraeus Kulzer GmbH, Hanau, Germany) were applied to the tooth surface using a disposable microbrush in a rubbing motion. After waiting for 30-60 seconds, the tooth surface was completely dried until the liquid disappeared and the surface lost its shine, and then rinsed with water.
  Other Names: Gluma Desensitizer
  Arms: Hydroxyethyl Methacrylate and Glutaraldehyde (Gluma)

SUMMARY:
The objective of this research was to evaluate the clinical success of desensitization treatments using four different materials in the first permanent molars (FPMs) affected by MIH.

DETAILED DESCRIPTION:
A total of 121 teeth with a Schiff cold air sensitivity scale (SCASS) score of 2 or 3 were included in 52 children (between 7-14 years). The FPMs were randomized into four groups; 5% sodium fluoride varnish (Group 1), silver diamine fluoride (Group 2), ammonia-free aqueous silver fluoride (Group 3), and hydroxyethyl methacrylate with glutaraldehyde (Group 4). Clinical evaluations were conducted at baseline, 15 minutes post-treatment, and at 1-week, 1-month, and 6-month follow-up. The two methods used at baseline for sensitivity assessment (SCASS for air sensitivity and the Wong-Baker pain rating scale for touch sensitivity) were used. Pain status during tooth brushing, pain during consumption of hot/cold/sweet/sour foods and beverages, pain during breathing (present/absent), gingival irritation, taste changes, post-eruptive breakdown, caries, spontaneous pain, mucosal swelling/fistula tract, mobility, and percussion/palpation sensitivity were evaluated. All sensitivity assessments were performed blindly by a researcher who did not know the baseline scores or the treatment administered. Statistical analysis was performed using SPSS 27.0 software (IBM Corp., Chicago, IL, USA) and the level of significance was set at p<0.05. The assumption of normal distribution was checked using the Shapiro-Wilk test. The Kruskal-Wallis test was used to compare three or more independent groups that did not have a normal distribution. The Friedman test was performed to examine the difference between three dependent groups where the normality assumption was not met. Post Hoc Adjusted Bonferroni tests were performed to determine the group or groups causing the difference. To test the relationship between categorical variables, the Pearson chi-square test was applied when the sample size assumption (expected value >5) was met, and Fisher's exact chi-square test was applied when the sample size assumption was not met.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children, aged 7-14 years, who attended the pediatric dentistry clinic regular dental examination
* Cooperative children diagnosed with MIH according to European Academy of Paediatric Dentistry (EAPD) criteria
* Presenting at least one FPMs that were fully erupted and has level 2 or 3 according to the Schiff Cold Air Sensitivity Scale

Exclusion Criteria:

* Children having hypomineralized FPMs with post-eruptive breakdown, cavitated carious lesions, restorations or fixed orthodontic appliances
* Enamel defect due to a condition other than MIH
* FPMs to be treated must not have been previously treated with a desensitizing agent.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Schiff Cold Air Sensitivity Scale for air sensitivity | 6 months
  Clinical evaluations were conducted at baseline, 15 minutes post-treatment, and at 1-week, 1-month, and 6-month follow-up. The The Schiff Cold Air Sensitivity Scale (SCASS) was used by the examiner to assess the subjects' response to this stimulus. Scoring was performed as follows: 0=subject does not respond to air stimulus; 1=subject responds to air stimulus but does not request discontinuation of stimulus; 2=subject responds to air stimulus and requests discontinuation or moves away from stimulus; and 3=subject responds to air stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
Wong-Baker Pain Rating Scale for tactile sensitivity | 6 months
  Clinical evaluations were conducted at baseline, 15 minutes post-treatment, and at 1-week, 1-month, and 6-month follow-up. Tactile hypersensitivity was assessed by scratching on the surface of the MIH-affected tooth with a dental explorer (max. twice scratches back and forth). The children scored pain intensity with the Wong Baker Faces Scale (WBFS) (0 = no hurt and 10 = hurts worst).

SECONDARY OUTCOMES:
Hypersensitivity during tooth brushing, consumption of hot/cold/sweet/sour foods and beverages or during breathing | 6 months
  Clinical evaluations were conducted at baseline, 15 minutes post-treatment, and at 1-week, 1-month, and 6-month follow-up. Pain status during tooth brushing, pain during consumption of hot/cold/sweet/sour foods and beverages, pain during breathing (present/absent), gingival irritation, taste changes, post-eruptive breakdown, caries, spontaneous pain, mucosal swelling/fistula tract, mobility, and percussion/palpation sensitivity were evaluated (present/absent).

CONTACTS AND LOCATIONS:
Overall Officials: Beste Ozgur, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozgul BM, Saat S, Sonmez H, Oz FT. Clinical evaluation of desensitizing treatment for incisor teeth affected by molar-incisor hypomineralization. J Clin Pediatr Dent. 2013 Winter;38(2):101-5. PMID 24683770
- [Background] Cavalcante BGN, Mlinko E, Szabo B, Teutsch B, Hegyi P, Vag J, Nemeth O, Gerber G, Varga G. Non-Invasive Strategies for Remineralization and Hypersensitivity Management in Molar-Incisor Hypomineralization-A Systematic Review and Meta-Analysis. J Clin Med. 2024 Nov 26;13(23):7154. doi: 10.3390/jcm13237154. PMID 39685613
- [Background] Ballikaya E, Unverdi GE, Cehreli ZC. Management of initial carious lesions of hypomineralized molars (MIH) with silver diamine fluoride or silver-modified atraumatic restorative treatment (SMART): 1-year results of a prospective, randomized clinical trial. Clin Oral Investig. 2022 Feb;26(2):2197-2205. doi: 10.1007/s00784-021-04236-5. Epub 2021 Nov 6. PMID 34743243
- [Background] Weerheijm KL, Jalevik B, Alaluusua S. Molar-incisor hypomineralisation. Caries Res. 2001 Sep-Oct;35(5):390-1. doi: 10.1159/000047479. No abstract available. PMID 11641576